CLINICAL TRIAL: NCT05673486
Title: Analgesic Efficacy of Regional Anesthesia by PENG-Block in Patients Diagnosed With Hip Fractures in the Emergency Department: an Open-label Randomized Controlled Trial
Brief Title: Regional Anesthesia by PENG-Block in Emergency Department
Acronym: ED-PENGBLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-CHITS-011; 2022-A02203-40 (Other: Id-RCB)
Record Dates: First submitted 2023-01-02; First posted 2023-01-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures
Keywords: Regional anesthesia; PENG block; Morphine consumption; Opioid sparing; Multimodal analgesia; Femoral neck fracture, intertrochanteric region fracture; Emergency department; Emergency medicine physician
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block + multimodal IV analgesia (Experimental): PENG block + multimodal IV analgesia (Nefopam, Paracetamol, Morphine)
  Interventions: Combination Product: PENG Block; Combination Product: Multimodal analgesia
- Multimodal analgesia alone (Active Comparator): Multimodal IV analgesia (Nefopam, Paracetamol, Morphine)
  Interventions: Combination Product: Multimodal analgesia

INTERVENTIONS:
Combination Product: PENG Block — With the patient in the supine position, the ultrasound probe is placed on a transverse plane over the anterior superior iliac spine (ASIS). Once the ASIS is identified, the transducer is aligned with the pubic ramus and rotated at approximately 45 degrees, parallel to the inguinal crease. The transducer is then slid medially along this axis until the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), and the psoas tendon is clearly identified, serving as anatomic landmarks.
  Sliding the probe distally or gently tilting the caudal will expose the head of the femur. Returning to the initial starting position, a needle is inserted in-plane, from lateral to medial, in the plane between the psoas tendon and the pubic ramus. 100 mg of ropivacaine is then deposited in this plane, lifting the psoas tendon.
  Arms: PENG block + multimodal IV analgesia
Combination Product: Multimodal analgesia — Multimodal analgesia is administered to patients as follows : 2-3 mg of morphine (2mg if patient's weight <60kg; 3mg if patient's weight >60kg) + Paracetamol 1g/8h and Nefopam 20mg/8h. Frequency of morphine administration depends on the assessed pain.

SUMMARY:
The study is a single-centre, open-label randomized comparative trial. Adult patients admitted to the emergency department for a hip fracture will be enrolled.

Pericapsular nerve block (PENG-block) is a regional anesthesia technique developed primarily as an analgesic technique in a perioperative setting during hip fractures related surgical procedures. Some authors propose the use of PENG-Block as an alternative to fascia iliaca block and femoral block for the analgesic management of hip fracture in the emergency department, but scientific evidence is weak in this setting.

The hypothesis of this study is that the use of PENG Block in the emergency department provides a better pain management for patients suffering from hip fractures with less opioid use.

DETAILED DESCRIPTION:
Pericapsular nerve block (PENG-block) is a regional anesthesia technique first described in 2018 and developed primarily as an analgesic technique in a perioperative setting during hip fractures related surgical procedures. The analgesic treatment with PENG-Block prevents motor block and thus reduces risk of intra-hospital falls. It also allows patients to get back on their feet more quickly and thus reduces loss of autonomy and risk of dependency. Moreover, it is a technique with a good safety profile that appears to be appropriate, feasible and effective in the context of the analgesic management of hip fractures in the emergency department. Therefore, some authors propose the use of PENG Block as an alternative to fascia iliaca block and femoral block for the analgesic management of this type of fracture.

The main objective of this study is to evaluate the effect of PENG Block combined with conventional multimodal analgesia when compared with conventional multimodal analgesia alone in terms of reduction of total morphine consumption in patients admitted to the emergency department for a hip fracture. The primary endpoint is the total morphine consumption from admission up to 24 hours after randomization or until surgery if the patient is operated on before 24 hours. The secondary objectives are : to assess whether the use of PENG-Block has an influence on the pain felt by the patient compared to conventional analgesia alone; to describe the tolerance of analgesia in the 2 groups; to assess whether the use of PENG-Block has an influence on the duration of hospitalization in the emergency department compared to conventional analgesia alone.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old) admitted to the emergency department for a hip fracture
2. Pain assessed by VAS/NRS ≥ 3 when the clinical suspicion of hip fracture is confirmed by the emergency physician
3. Patients capable of expressing his/her consent prior to participation in the study
4. Affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

1. Patients for who it is impossible to collect the pain assessment scale
2. Patients with known or suspected bleeding disorders :

   * Personal and family history of bleeding symptoms (spontaneous or induced)
   * Clinical signs suggesting a haemostasis disorder
   * Patient on anticoagulant at a curative dose with a very high risk of bleeding (labile International Normalized Ratio (INR), mechanical valve, acute kidney failure and treatment with direct oral anticoagulants)
   * Inherited bleeding disorder (Hemophilia A, Hemophilia B, Von Willebrand disease, Fibrinogen deficiency, Factor XII deficiency)
   * Pathologies that may interfere with hemostasis: advanced liver disease, decompensated hematological disease, collagen diseases such as Ehlers-Danlos disease
3. Patients in whom it is impossible to perform the PENG-Block: Body Mass Index (BMI) > 40, adenopathy or infection at the puncture site, allergy to the anesthetics used
4. Pregnant, parturient or breastfeeding women
5. Patients under judicial protection or judicial safeguard
6. Any other reason which, in the opinion of the investigator, could interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | Up to 24 hours after randomization
  Total morphine consumption in mg per hour from admission up to 24 hours after randomization or until surgery if the patient is operated on before 24 hours

SECONDARY OUTCOMES:
Pain intensity according to a Numeric Rating Scale (NRS) | Up to 24 hours after randomization
  The patient's pain will be assessed using a Numeric Rating Scale at the start of care in the emergency department, when the clinical suspicion of hip fracture is confirmed by the emergency doctor, then every hour in the emergency room and every 4 hours in the surgery department for 24 hours or until transfer to the operating room if the surgery takes place before.
  The minimum value of the scale, corresponding to no pain at all, is 0 and the maximum value is 10.
Presence of side effects | Up to 24 hours after randomization
  The tolerance of analgesic treatments will be assessed by evaluating the presence or absence of side effects, during the first 24 hours of treatment or until surgery if it takes place before :
  Side effects related to opioids such as Confusion, Bradypnea, Nausea or vomiting Side effects related to PENG-Block such as Pain at the puncture site, Acute retention of urine, Bleeding Any other adverse effects occurring during the study will be collected.
Duration of hospitalization in the emergency department | Up to 24 hours after randomization
  Duration of care in hours at the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent CAUMON, MD, Study Director — Centre Hospitalier de Hyères
Locations (1):
- Hyères Hospital, Hyères, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calati P, Lenoir C, Kamel LC, Contie N, Firoloni JD, Sichez A, Sebai A, Chelly J, Caumon L. Effectiveness of pericapsular nerve group block for hip fracture pain management in the emergency department: results of the ED-PENG-B randomised controlled trial. BMC Emerg Med. 2025 Nov 26;25(1):245. doi: 10.1186/s12873-025-01401-x. PMID 41299315